CLINICAL TRIAL: NCT01118182
Title: Use of a Traumatic Brain Injury (TBI) Screen in a Veteran Mental Health Population: Prevalence, Validation, and Psychiatric Outcomes
Brief Title: Use of a Traumatic Brain Injury (TBI) Screen in a Veteran Mental Health Population
Acronym: TBI
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: Colorado Traumatic Brain Injury Trust Fund (Other); Ohio State University (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Lisa Brenner, Director, VA VISN 19 Mental Illness Research Education and Clinical Center (MIRECC), VA Eastern Colorado Health Care System
Other Study IDs: COMIRB08-0001
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Veterans; Psychiatric Disorders; Suicide
MeSH Terms: conditions — Brain Injuries, Traumatic; Mental Disorders; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traumatic Brain Injury (TBI): Veterans with a positive history of TBI
- No Traumatic Brain Injury (TBI): Veterans with a negative history of TBI

SUMMARY:
The primary aims of this study are to: 1) Establish the concurrent criterion-related validity of four traumatic brain injury (TBI) screening questions (TBI-4) using the Ohio State University TBI Identification Method (OSU TBI-ID) and 2) Establish the concurrent criterion-related validity of the TBI-4 with the addition of detailed information elicited by the four questions. Secondary aims include: 1) Determining if the addition of detailed information elicited by the TBI-4 results in increased specificity; 2) Determining whether the prevalence of traumatic brain injury (TBI) in this sample is concordant with previous research; and 3) Determining whether psychiatric outcomes are worse for veterans with traumatic brain injury (TBI) than those with no traumatic brain injury(TBI).

DETAILED DESCRIPTION:
The primary aims of this study are to: 1) Establish the concurrent criterion-related validity of four traumatic brain injury (TBI) screening questions (TBI-4) using the Ohio State University TBI Identification Method (OSU TBI-ID) and 2) Establish the concurrent criterion-related validity of the TBI-4 with the addition of detailed information elicited by the four questions. Secondary aims include: 1) Determining if the addition of detailed information elicited by the TBI-4 results in increased specificity; 2) Determining whether the prevalence of traumatic brain injury (TBI) in this sample is concordant with previous research; and 3) Determining whether psychiatric outcomes are worse for veterans with traumatic brain injury (TBI) than those with no traumatic brain injury(TBI).

Primary Hypotheses:

Hypothesis 1a: The sensitivity and specificity of the TBI-4 will be significantly greater than 0.75 and 0.80, respectively.

Hypothesis 1b: The sensitivity and specificity of the TBI-4 with the addition of detailed information elicited by these questions (i.e., free text information entered by the clinician who administered the TBI-4) will be significantly greater than 0.75 and 0.80, respectively.

Secondary Hypotheses:

Hypothesis 1c: The specificity of the TBI-4 with the addition of detailed information elicited by these questions (i.e., free text information entered by the clinician who administered the TBI-4) will be significantly greater than that of the four questions alone.

Hypothesis 2: A significant difference in psychiatric outcomes (psychiatric hospitalizations, suicidal ideation, suicide attempts and completions, and mental health-related contacts) will be identified in those with a history of TBI versus those without a history of TBI as determined, first, by the TBI-4 and, second, by the OSU TBI-ID.

Hypothesis 3: The prevalence of Traumatic Brain Injury- Loss of Consciousness (TBI-LOC) in this population will be similar to that identified by Walker et al1 (31.7% of individuals will report 1 or more TBI-LOC).

ELIGIBILITY:
Inclusion Criteria:

* Veteran must be at least 18 years of age.
* Veteran must have had a mental health intake no earlier than January of 2007.

Exclusion Criteria:

* Failure to provide informed consent as evidenced by inability to respond to the above stated questions.
* No Mental Health Intake note in the medical record.
* Presence of a Mental Health Intake note in the computer which does not contain the TBI-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indivduals with a history of completing the 4 Traumatic Brain Injury (TBI) screening questions during a mental health intake.
Sampling Method: Non-Probability Sample
Enrollment: 1810 (Actual)
Dates: Start 2009-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Ohio State University TBI Identification Method (OSU TBI-ID) | 1 day
  Structured clinical interview used as the gold standard for establishing a lifetime history of TBI

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — VISN 19 MIRECC
Locations (1):
- Denver VA Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Rocky Mountain MIRECC website — https://www.mirecc.va.gov/mirecc/visn19/